CLINICAL TRIAL: NCT00840788
Title: Skin Adhesive Versus Subcuticular Suture for Perineal Skin Repair After Episiotomy - a Randomized Controlled Trial.
Brief Title: Comparison of Adhesive Glue With Skin Suture for Repair of Episiotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Joao (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Diogo Ayres de Campos, Servico de Ginecologia e Obstetricia, Hospital de S. Joao
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Episio- 01 - RCT
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Mediolateral Episiotomy After Delivery
Keywords: skin adhesive; tissue adhesive; mediolateral episiotomy; perineal repair; labor and delivery; repair
MeSH Terms: interventions — octyl 2-cyanoacrylate; Polyglactin 910

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin adhesive (Experimental): perineal skin repair with octyl-2-cyanoacrylate skin adhesive
  Interventions: Procedure: octyl-2-cyanoacrylate adhesive glue
- subcuticular suture (Active Comparator): continuous subcuticular suture of perineal skin using rapidly absorbable polyglactin 910
  Interventions: Procedure: Subcuticular suture of perineal skin

INTERVENTIONS:
Procedure: octyl-2-cyanoacrylate adhesive glue — use of octyl-2-cyanoacrylate adhesive glue for perineal skin repair after episiotomy
  Other Names: Dermabond
  Arms: Skin adhesive
Procedure: Subcuticular suture of perineal skin — Use of continuous subcuticular suture with rapidly absorbable polyglactin 910 for closure of the perineal skin in episiotomy repair
  Other Names: Vicryl
  Arms: subcuticular suture

SUMMARY:
Surgical repair of perineal lesions after delivery is frequently associated with pain and discomfort interfering with the normal activities of the puerperium. The aim of this study was to compare perineal skin repair after episiotomy with adhesive glue versus a subcuticular suture, regarding the incidence of pain and wound complications.

ELIGIBILITY:
Inclusion Criteria:

* vaginal delivery
* episiotomy performed
* no further perineal or vaginal lesions present

Exclusion Criteria:

* previously existing local infections or lesions
* body mass index > 35 (Kg/m2)
* severe pulmonary disease
* collagen disease
* known immunodeficiency
* diabetes mellitus
* immunosuppressive treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Self-assessed perineal pain | First 30 days after delivery

SECONDARY OUTCOMES:
Total time spent with repair of episiotomy | within 1 hour after birth
Pain during procedure | within 1 hour after birth
Difficulties reported during procedure | within 1 hour after birth
Number of sutures and adhesive devices used | within 1 hour after birth
Wound complications | 42-68 hours after delivery
Need to seek health facilities | 30 days after delivery
Return of sexual activity | 30 days after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Diogo Ayres-de-Campos, PhD, Principal Investigator — Hospital de S. Joao, Faculdade de Medicina da Universidade do Porto
Locations (1):
- Servico de Ginecologia e Obstetricia, Hospital de S, Joao, Porto, Porto District, Portugal